CLINICAL TRIAL: NCT01040013
Title: GUT OXYGENATION DURING AND AFTER LAPAROSCOPIC AND OPEN COLON RESECTION. A RANDOMIZAD CLINICAL TRIAL
Brief Title: Gut Oxygenation and Laparoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: LUCA GIANOTTI, MD,SCD, MILNO-BICOCCA UNIVERSITY
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oxylap-2009
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2009-11

CONDITIONS: Laparoscopy; Laparotomy; Oxygenation,; Ischemia-Reperfusion Injury
Keywords: LAPAROSCOPY,; LAPAROTOMY,; OXYGENATION,; ISCHEMIA-REPERFUSION INJURY
MeSH Terms: conditions — Reperfusion Injury | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopy (Experimental): Laparoscopic Left-Sided Colectomy
  Interventions: Procedure: Laparoscopy
- laparotomy (Active Comparator): Laparotomic Left-Sided Colectomy
  Interventions: Procedure: left colectomy by laparotomy

INTERVENTIONS:
Procedure: Laparoscopy — Laparoscopic Left-Colectomy
  Arms: Laparoscopy
Procedure: left colectomy by laparotomy — PatientS will be operated by laparotomy
  Arms: laparotomy

SUMMARY:
Patients with left-colon cancer will be randomized to laparoscopic or laparotomic operation. during surgery and for 6 days after operation, intestinal oxygen tension and ischemia-reperfusion injury markers will be evaluated to understand if pneumoperitoneum is associated with reduced splanchnic blood flow and ischemia-reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Proven Cleft Colon Cancer, Signed Informed Consent

Exclusion Criteria:

* Emergency surgery,
* Cancer infiltrating adjacent organ (at CT scan),
* Severe cardiovascular (New York Heart Association class > 3 ),
* Respiratory (arterial PO2 < 70 mmHg),
* Renal (plasma creatinine > 3 MG/dL) or hepatic (Child C) dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Intestinal oxygenation | 7 DAYS

SECONDARY OUTCOMES:
Ischemic reperfusion injury | 7 DAYS

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gianotti, MD, PhD, Principal Investigator — Milano-Bicocca university
Locations (1):
- San Gerardo Hospital, Monza, Italy

REFERENCES:
- [Background] Moore K, Roberts LJ 2nd. Measurement of lipid peroxidation. Free Radic Res. 1998 Jun;28(6):659-71. doi: 10.3109/10715769809065821. PMID 9736317
- [Derived] Gianotti L, Nespoli L, Rocchetti S, Vignali A, Nespoli A, Braga M. Gut oxygenation and oxidative damage during and after laparoscopic and open left-sided colon resection: a prospective, randomized, controlled clinical trial. Surg Endosc. 2011 Jun;25(6):1835-43. doi: 10.1007/s00464-010-1475-2. Epub 2010 Dec 7. PMID 21136109